CLINICAL TRIAL: NCT00093756
Title: Phase I/II Study of PS-341 in Combination With Paclitaxel, Carboplatin, and Concurrent Thoracic Radiation Therapy for Non-small Cell Lung Cancer (NSCLC)
Brief Title: Bortezomib, Paclitaxel, Carboplatin and Radiation Therapy for Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00643; NCI-2009-00643 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000390108; NCCTG-N0321; N0321 (Other: North Central Cancer Treatment Group); N0321 (Other: CTEP); U10CA025224 (NIH)
Record Dates: First submitted 2004-10-06; First posted 2004-10-08 (Estimated); Results first posted 2014-12-08 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-11

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIA Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy, Conformal; Bortezomib; Paclitaxel; Carboplatin

ARMS (1):
- Treatment (bortezomib, paclitaxel, carboplatin) (Experimental): PHASE I: Cohorts of 3-6 patients receive escalating doses of study medications until the maximum tolerated dose (MTD) is determined. PHASE II: Patients receive as in phase I at the MTD. Patients also undergo radiotherapy as in phase I.
  3-dimensional conformal radiation therapy bortezomib: Given IV paclitaxel: Given IV carboplatin: Given IV
  Interventions: Radiation: 3-dimensional conformal radiation therapy; Drug: bortezomib; Drug: paclitaxel; Drug: carboplatin

INTERVENTIONS:
Radiation: 3-dimensional conformal radiation therapy
Drug: bortezomib — Given IV
Drug: paclitaxel — Given IV
Drug: carboplatin — Given IV

SUMMARY:
This phase I/II trial (phase I closed to accrual as of 09/29/2009) is studying the side effects and best dose of bortezomib, paclitaxel, and carboplatin when given with radiation therapy and to see how well they work in treating patients with stage IIIA or stage IIIB non-small cell lung cancer that cannot be removed by surgery. Bortezomib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Drugs used in chemotherapy, such as paclitaxel and carboplatin, work in different ways to stop tumor cells from dividing so they stop growing or die. Bortezomib may increase the effectiveness of paclitaxel and carboplatin by making tumor cells more sensitive to the drugs. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving bortezomib, paclitaxel, and carboplatin together with radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of bortezomib, paclitaxel, and carboplatin when administered with fractionated radiotherapy in patients with unresectable stage IIIA or IIIB non-small cell lung cancer. (Phase I) (closed to accrual as of 09/29/2009) II. Determine the 1-year survival of patients treated with this regimen. (Phase II)

SECONDARY OBJECTIVES:

I. Determine the tolerability of this regimen in these patients. (Phase II) II. Determine the response rate, progression-free survival, and overall survival of patients treated with this regimen. (Phase II) III. Correlate p27 expression in tumor tissue with survival, time to progression, and response in patients treated with this regimen. (Phase II)

OUTLINE: This is a multicenter, phase I (closed to accrual as of 09/29/2009), dose-escalation study of bortezomib, paclitaxel, and carboplatin followed by a phase II study.

PHASE I: (closed to accrual as of 09/29/2009) Patients receive bortezomib IV on days 1, 4, 8, and 11. Patients also receive paclitaxel IV over 3 hours followed by carboplatin IV over 30 minutes on day 2. Patients undergo radiotherapy once daily on days 1-5, 8-12, 15-19. Treatment repeats every 3 weeks up to 2 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of bortezomib, paclitaxel, and carboplatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

PHASE II: Patients receive bortezomib, paclitaxel, and carboplatin as in phase I at the MTD. Patients also undergo radiotherapy as in phase I. Patients are followed up periodically for up to 5 years from the time of registration.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer (NSCLC)
* Locally advanced stage IIIA or IIIB disease that is considered unresectable
* No stage IV disease
* Requires radiotherapy
* Performance status (PS) - Eastern Cooperative Oncology Group (ECOG) 0-1
* At least 12 weeks
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* aspartate aminotransferase (AST) ≤ 3 times ULN
* Creatinine ≤ 1.5 times ULN
* No New York Heart Association class III or IV heart disease
* Forced expiratory volume (FEV) FEV_1 ≥ 1 L OR 35% of predicted
* Weight loss < 10% within the past 3 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No peripheral neuropathy ≥ grade 2
* No other severe underlying disease that would preclude study participation
* No uncontrolled infection
* No unhealed wound within the past 2 weeks
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, adequately treated noninvasive carcinomas (carcinoma in situ), or localized prostate cancer
* No concurrent prophylactic filgrastim (G-CSF) or sargramostim (GM-CSF)
* No prior systemic chemotherapy for NSCLC*
* No prior radiotherapy to the chest
* More than 2 weeks since prior major surgery

Contraindications

* Any of the following:

  * Pregnant wome
  * Nursing women
  * Men or women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], or abstinence, etc.) as this regimen may be harmful to a developing fetus or nursing child NOTE: This study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown.
* Any of the following prior therapies:

  * Prior radiation therapy to the chest
  * Prior systemic chemotherapy for NSCLC (phase II portion)
* New York Heart Association classification III or IV (see Appendix II).
* Any other severe underlying diseases which are, in the judgment of the investigator, inappropriate for entry into this study.
* uncontrolled infection.
* Major surgery or unhealed wound ≤ 2 weeks prior to registration.
* Prior history of malignancy ≤ 5 years, except for adequately treated basal cell or squamous cell skin cancer, adequately treated noninvasive carcinomas (carcinoma in situ), or localized prostate cancer.
* Peripheral neuropathy ≥grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-09; Primary Completion 2012-01 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alex Adjei, Principal Investigator — North Central Cancer Treatment Group
Locations (143):
- United States (143):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Saint Anthony Memorial Hospital, Effingham, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Holy Family Medical Center, Monmouth, Illinois
  - Illinois CancerCare-Monmouth, Monmouth, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Community Cancer Center, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - OSF Saint Francis Medical Center Radiation Oncology Service at the Central Illinois Comprehensive CC, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare-Spring Valley, Spring Valley, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Carle Foundation - Carle Cancer Center, Urbana, Illinois
  - Saint Anthony Memorial Health Center, Michigan City, Indiana
  - Saint Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Harris, John Gilbert MD (UIA Investigator), Alexandria, Minnesota
  - Brainerd Medical Center Inc, Brainerd, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Duluth Clinic CCOP, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Adult and Pediatric Urology PLLP, Sartell, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Geisinger Medical Center, Danville, Pennsylvania
  - Geisinger Medical Center-Cancer Center Hazelton, Hazleton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - AnMed Health Hospital, Anderson, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Upstate Carolina CCOP, Spartanburg, South Carolina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fifty two (52) patients were accrued, out of which 4 were cancels. Twenty one (21) patients were accrued for phase I portion of the study. Twenty Seven (27) patients are accrued for phase II portion of the study. Twenty Seven (27) Phase II patients are evaluable for primary outcome measure.
Groups:
- Phase I: PHASE I: Cohorts of 3-6 patients receive escalating doses of study medications until the maximum tolerated dose (MTD) is determined. 3-dimensional conformal radiation therapy, bortezomib: Given IV, paclitaxel: Given IV, carboplatin: Given IV.
- Phase II: PHASE II: Patients receive as in phase I at the MTD. Patients also undergo radiotherapy as in phase I. 3-dimensional conformal radiation therapy, bortezomib: Given IV, paclitaxel: Given IV, , carboplatin: Given IV.
Period: Overall Study
Arm/Group | Phase I | Phase II
Started | 27 | 21
Completed | 27 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PhaseI: PHASE I: Cohorts of 3-6 patients receive escalating doses of study medications until the maximum tolerated dose (MTD) is determined. 3-dimensional conformal radiation therapy> bortezomib: Given IV> paclitaxel: Given IV> carboplatin: Given IV
- PhaseII: PHASE II: Patients receive as in phase I at the MTD. Patients also undergo radiotherapy as in phase I. 3-dimensional conformal radiation therapy> bortezomib: Given IV> paclitaxel: Given IV> carboplatin: Given IV
- Total: Total of all reporting groups
Arm/Group | PhaseI | PhaseII | Total
Number analyzed (Participants) | 27 | 21 | 48
Age, Continuous [Median (Full Range); unit: years] | 63 [45 to 78] | 58 [43 to 79] | 58 [43 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 17 | 13 | 30
Region of Enrollment [Number; unit: participants]
  United States | 21 | 27 | 48

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint of This Trial is the Proportion of Patients Alive at 1 Year. Phase II Patients Only.
Description: The primary endpoint of this trial is the proportion of patients alive at 1 year (i.e., 365 days) after study registration. Proportion of successes, defined as the number of patients alive at one year divided by the total number of evaluable patients.
Time Frame: At 1 year
Population: This analysis included all 21 patients enrolled in the Phase II portion of the study and 6 patients enrolled in the Phase I who were treated at the Phase II dose level.
Measure: Number; unit: proportion of Participants
Groups:
- PhaseII: PHASE II: Patients receive as in phase I at the MTD. Patients also undergo radiotherapy as in phase I. 3-dimensional conformal radiation therapy, bortezomib: Given IV, paclitaxel: Given IV, carboplatin: Given IV.
Arm/Group | PhaseII
Number analyzed (Participants) | 27
proportion of Participants | 0.73

2. Secondary Outcome: Confirmed Tumor Response
Description: Response was assessed using the RECIST v1.1 criteria. Patients were evaluated at 4 weeks post-RT, 3 months post-RT, every 3 months for 1 year post-RT, and every 6 months thereafter for a maximum of 5 years from time of registration. A Complete Response (CR) is defined as the disappearance of all target lesions. A Partial Response (PR) is defined as at least a 20% decrease in the sum of the longest diameter of target lesions from baseline. A confirmed response is defined as a CR or PR as the objective status on 2 consecutive evaluations at least 4 weeks apart.
Time Frame: Up to 5 years
Population: All 21 patients from Phase II and 6 patients registered to the Phase II dose level of Phase I were included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- PhaseII: PHASE II: Patients receive as in phase I at the MTD. Patients also undergo radiotherapy as in phase I. 3-dimensional conformal radiation therapy, bortezomib: Given IV, paclitaxel: Given IV, , carboplatin: Given IV.
Arm/Group | PhaseII
Number analyzed (Participants) | 27
Participants
  Complete Response (CR) | 3
  Partial Response (PR) | 4

3. Secondary Outcome: Time to Progression
Description: The distribution of time to progression will be estimated using the method of Kaplan-Meier.
Time Frame: From study registration to date of disease progression or date of last follow-up, up to 5 years
Population: Study team decision not to run this analysis.
Groups:
- Phase II: PHASE II: Patients receive as in phase I at the MTD. Patients also undergo radiotherapy as in phase I. 3-dimensional conformal radiation therapy, bortezomib: Given IV, paclitaxel: Given IV, carboplatin: Given IV.
Arm/Group | Phase II
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-free Survival
Description: The distribution of progression-free survival (PFS) is defined as the time from registration to the time of progression or death, whichever comes first. The PFS will be estimated using the method of Kaplan-Meier.
Time Frame: From study registration to the first of either death due to any cause or progression, up to 5 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 27
months | 8.4 [4.1 to 10.5]

5. Secondary Outcome: Overall Survival
Description: Overall Survival is defined as the time from registration to the time to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: From registration to death due to any cause, up to 5 years
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 27
months | 25 [15.6 to 35.8]

6. Secondary Outcome: Frequency and Severity of Observed Toxicity, Graded by Common Terminology Criteria for Adverse Events (CTCAE)
Description: Toxicity was reported after the first 21 days of treatment and after each 28 day cycle thereafter. Events were graded according to the Common Terminology Criteria for Adverse Events (CTCAE) v3.0. The number of patients reporting grade 3 and higher are tabulated.
Time Frame: Up to 5 years
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II
Number analyzed (Participants) | 27
Participants
  Grade 3 Adverse Event | 22
  Grade 4 Adverse Event | 15

ADVERSE EVENTS:
Groups:
- PhaseI: PHASE I: Cohorts of 3-6 patients receive escalating doses of study medications until the maximum tolerated dose (MTD) is determined. 3-dimensional conformal radiation therapy, bortezomib: Given IV, paclitaxel: Given IV, carboplatin: Given IV.
Arm/Group | PhaseI | PhaseII
Serious Adverse Events (participants affected / at risk) | 9/21 | 12/27
Other Adverse Events (participants affected / at risk) | 21/21 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PhaseI (N=21) | PhaseII (N=27)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischemia (Cardiac disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 1 (1) | 5 (5)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 6 (6)
Platelet count decreased (Investigations) | 0 (0) | 9 (9)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum phosphate decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 1 (1) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PhaseI (N=21) | PhaseII (N=27)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 17 (36) | 23 (64)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 4 (5) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 11 (15) | 9 (16)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 17 (42) | 21 (40)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 6 (9) | 7 (8)
Esophageal mucositis (Gastrointestinal disorders) | 6 (8) | 13 (17)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 1 (2)
Mucositis oral (Gastrointestinal disorders) | 5 (8) | 9 (13)
Nausea (Gastrointestinal disorders) | 15 (24) | 21 (35)
Vomiting (Gastrointestinal disorders) | 7 (10) | 12 (18)
Chest pain (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 20 (60) | 26 (68)
Fever (General disorders) | 4 (4) | 4 (5)
Pain (General disorders) | 1 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
Gingival infection (Infections and infestations) | 1 (1) | 1 (1)
Paranasal sinus infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 10 (14) | 14 (21)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
INR increased (Investigations) | 1 (2) | 0 (0)
Leukocyte count decreased (Investigations) | 19 (36) | 22 (43)
Lymphocyte count decreased (Investigations) | 3 (4) | 1 (1)
Neutrophil count decreased (Investigations) | 17 (24) | 20 (34)
Platelet count decreased (Investigations) | 13 (19) | 23 (31)
Weight loss (Investigations) | 1 (1) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 4 (4)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Serum albumin decreased (Metabolism and nutrition disorders) | 1 (2) | 1 (2)
Serum calcium decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Serum magnesium decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (10) | 12 (27)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (2)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 1 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 11 (27) | 15 (38)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (51) | 21 (45)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (5) | 9 (13)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 3 (4) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less